CLINICAL TRIAL: NCT01555307
Title: Effectiveness of Exercise Programs Following Total Hip and Knee Joint Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-06-461; 12697E (Other: REB)
Record Dates: First submitted 2012-01-16; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-01

CONDITIONS: Hip and Knee Joint Osteoarthritis; Hip and Knee Joint Arthroplasty
Keywords: total hip arthroplasty; total knee arthroplasty; balance exercises; force plate; berg balance scale; timed up and go test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance group (Experimental): Typical plus balance exercises
  Interventions: Other: Typical range of motion and muscle strengthening exercises, and balance exercises
- Typical group (Other): Typical exercises
  Interventions: Other: Typical group

INTERVENTIONS:
Other: Typical range of motion and muscle strengthening exercises, and balance exercises — Seven typical exercises, and three balance exercises, 10 times each, 3 times a day.
  Arms: Balance group
Other: Typical group — Seven typical exercises, 10 times each, 3 times a day
  Arms: Typical group

SUMMARY:
The purpose of the study was to evaluate the effectiveness of balance exercises added to typical joint range of motion and muscle strengthening exercises on balance in patients following total hip or knee joint arthroplasty

DETAILED DESCRIPTION:
Rehabilitation program following total hip and knee joint arthroplasty typically focus on joint range of motion and muscle strengthening exercises. Although the balance ability of these patients tends to be reduced, leading to limitations in mobility and activities of daily living, clinicians often assume that strength and joint range of motion exercises will ultimately lead to improvement in balance, making the typical exercise programs appropriate. However, the feasibility and effectiveness of introducing balance specific exercises during the post-operative period is unclear.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary unilateral total hip or knee joint arthroplasty.
* Patients who had been advised to weight bear as tolerated following surgery.

Exclusion Criteria:

* Patients who had been advised by their surgeon to remain non-weight bearing or partial weight bearing on the operated leg or unoperated leg.
* Patients with neurological conditions such as hemiplegia, peripheral neuropathy, Parkinsons disease, multiple sclerosis, or spinal cord compression that might affect balance.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | Day 0 and Week 5

SECONDARY OUTCOMES:
Timed Up and go test | Day 0 and Week 5
Western Ontario McMaster Universities Osteoarthritis Index | Day 0 and Week 5
Activity-specific Balance Confidence Scale | Day 0 and Week 5
Force platform | Week 5

CONTACTS AND LOCATIONS:
Overall Officials: John Kramer, PhD, Principal Investigator — Western University, Canada
Locations (1):
- School of Physical Therapy, University of Western Ontario, London, Ontario, Canada